CLINICAL TRIAL: NCT00292071
Title: A Multicenter, Open, Sequential Dose-Escalation Study to Investigate the Safety, Tolerability, and Pharmacokinetics of 2 Separate Doses of Caspofungin Acetate in Children Between the Ages of 3 to 24 Months With New Onset Fever and Neutropenia
Brief Title: Open, Pharmacokinetic Study of Caspofungin Acetate in Immunocompromised Young Children With Febrile Neutropenia (0991-042)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-042; MK0991-042; 2005_099
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Caspofungin

ARMS (2):
- 1 (Other): IV caspofungin acetate (50 mg/m²/day)
  Interventions: Drug: caspofungin acetate
- 2 (Other): IV caspofungin acetate (70 mg/m²/day)
  Interventions: Drug: caspofungin acetate

INTERVENTIONS:
Drug: caspofungin acetate — (50 mg/m²/day and 70 mg/m²/day) Caspofungin will be given for a minimum of 4 days (or at least 2 separate days of 7-point plasma sampling). Patients will be administered caspofungin for a maximum of 28 days.
  Other Names: MK0991; CANCIDAS®

SUMMARY:
This is an open-label study of MK0991 in children between 3 to 24 months of age with new onset fever and neutropenia. The purpose of the study is to investigate plasma drug levels of caspofungin.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 3 to 24 months of age with one or more of the following conditions:
* Leukemia, lymphoma, or other cancers
* Bone marrow or peripheral stem transplantation
* High dose chemotherapy leading to a decrease in white blood cells
* Aplastic anemia
* Patient has an absolute neutrophil count <500 mm3 (a specific type of white blood cell that fights infection) AND at least one recording of fever > 38 degreesC (oral or oral equivalent) within 72 hours of screening.

Exclusion Criteria:

* Patient is <3 months or >24 months of age at the time of study drug administration
* Patient has proven or probable invasive fungal infection at the time of enrollment
* Patient has certain blood clotting or liver function abnormalities
* Patient is hemodynamically unstable, exhibits hemodynamic compromise or is not expected to survive at least 5 days
* Patient is taking rifampin, cyclosporin A, phenytoin, carbamazepine, or phenobarbital.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2004-05; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Plasma drug-level observed in children 3 to 24 months of age is similar to the levels observed in adults. | 28 Days

SECONDARY OUTCOMES:
Caspofungin is generally safe and well tolerated in children 3 to 24 months of age. | 28 Days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Neely M, Jafri HS, Seibel N, Knapp K, Adamson PC, Bradshaw SK, Strohmaier KM, Sun P, Bi S, Dockendorf MF, Stone JA, Kartsonis NA. Pharmacokinetics and safety of caspofungin in older infants and toddlers. Antimicrob Agents Chemother. 2009 Apr;53(4):1450-6. doi: 10.1128/AAC.01027-08. Epub 2008 Dec 29. PMID 19114680
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html